CLINICAL TRIAL: NCT02989623
Title: A Pilot Phase I Open Label Study of Cu-64-TP3805 PET Imaging for Detection of Prostate Cancer in Men With Persistently Elevated PSA
Brief Title: Copper Cu 64 TP3805 PET in Detecting Prostate Cancer in Patients With Persistently Elevated PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15F.264; R01CA157372 (NIH); JT 7709 (Other: JeffTrial Number)
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2025-03-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (copper Cu 64 TP3805, PET/CT, biopsy) (Experimental): Patients receive copper Cu 64 TP3805 IV over 5 minutes and 30 minutes and 2 hours later, undergo whole body Positron Emission Tomography/Computed Tomography (PET/CT) imaging over 1 hour.
  Interventions: Radiation: Copper Cu 64 TP3805; Procedure: Positron Emission Tomography and Computed Tomography Scan

INTERVENTIONS:
Radiation: Copper Cu 64 TP3805 — Given Intravenously
  Other Names: Cu-64-TP3805
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo copper Cu 64 TP3805 PET/CT scan
  Other Names: PET/CT SCAN; Positron Emission Tomography/Computed Tomography

SUMMARY:
This pilot phase I trial studies how well copper Cu 64 TP3805 positron emission tomography (PET) works in detecting prostate cancer in patients with persistently elevated prostate specific antigen (PSA). The copper Cu 64 TP3805 PET scan uses copper Cu 64 TP3805, a compound made of a radioactive agent attached to a molecule that looks like a hormone that binds to cancer cells to detect prostate cancer during PET scans. Copper Cu 64 TP3805 PET may be able to see tumors at an earlier stage than the standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of Cu-64-TP3805 (copper Cu 64 TP3805) to detect prostate cancer (PC), or absence thereof, within the prostate gland.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed informed consent and willingness to comply with protocol requirements
* Persistently elevated PSA
* Scheduled for magnetic resonance imaging (MRI) fusion/transrectal ultrasound (TRUS) biopsy, followed by histology
* Agree to use an acceptable form of birth control for a period of 7 days after the Cu-64-TP3805 injection

Exclusion Criteria:

* Participating would significantly delay the scheduled standard of care therapy
* Administered a radioisotope within 10 physical half-lives prior to study drug injection
* Have any medical condition or other circumstances that, in the opinion of the investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Thakur, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Copper Cu 64 TP3805, PET/CT, Biopsy)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Copper Cu 64 TP3805, PET/CT, Biopsy)
Number analyzed (Participants) | 25
Age, Customized [Mean (Standard Deviation); unit: years] | 63.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Prostate Cancer Detection Within the Prostate Gland by Copper Cu 64 TP3805 PET
Description: The proportion of participants with lesions detected with copper Cu-64 PET will be determined with the lesion as the unit of analysis. 95% confidence intervals will be calculated.
Time Frame: At 3 weeks post imaging visit
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Copper Cu 64 TP3805, PET/CT, Biopsy)
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: Total Incidence of Multiple Lesions in an Individual Patient
Description: Generalized Estimating Equations will be utilized to provide a total number of lesions
Time Frame: At 3 weeks post imaging procedure
Measure: Number; unit: lesions
Arm/Group | Diagnostic (Copper Cu 64 TP3805, PET/CT, Biopsy)
Number analyzed (Participants) | 25
lesions | 339

ADVERSE EVENTS:
Time Frame: subjects were monitored for 24 hours post imaging for adverse events
Description: all adverse events were related to standard of care
Arm/Group | Diagnostic (Copper Cu 64 TP3805, PET/CT, Biopsy)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT02989623/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT02989623/ICF_001.pdf